CLINICAL TRIAL: NCT00079599
Title: Phase II Developmental Study on Fatigue in AIDS Patients
Brief Title: L-Carnitine to Treat Fatigue in AIDS Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Ricardo Cruciani, MD, PHD, Vice-Chairman, Department of Pain and Palliative Care, Director, Research Division, Beth Israel Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R21NR008295-01 (NIH)
Record Dates: First submitted 2004-03-09; First posted 2004-03-10 (Estimated); Last update posted 2008-09-04 (Estimated); Status verified 2008-09

CONDITIONS: HIV Infections; AIDS
Keywords: Carnitine Deficiency; Fatigue; Complementary Therapies
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Systemic carnitine deficiency; Fatigue | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: L-carnitine
- 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: L-carnitine — A study drug, L-carnitine, titrating the doses from 0.5 g to 3 g to reduce the possibility of side effects, lasting for two weeeks followed by an extension phase where all patients recieved L-carnitine for an additional two weeks.
  Arms: 1
Other: Placebo — A placebo, where patients underwent the dose titration identical to the study patients, lasting for two weeeks followed by an extension phase where all patients recieved L-carnitine for an additional two weeks.
  Arms: 2

SUMMARY:
Patients with AIDS may develop a deficiency of the micronutrient carnitine and such a deficiency may contribute to fatigue in these patients. This study will determine whether carnitine supplementation will improve fatigue and related symptoms in carnitine-deficient patients with AIDS.

DETAILED DESCRIPTION:
Fatigue is a commonly reported symptom in patients with end stage AIDS. Appropriate treatment can relieve suffering and improve quality of life. The role of progression of the disease, depression, anemia, and poor nutritional status in the development of fatigue is well recognized. However, the impact of micronutrient deficiencies has been minimally explored. AIDS patients are at risk for micronutrient deficiencies because of decreased caloric intake, increased metabolic requirements, and treatment with medications that can interfere with absorption, synthesis, and excretion. Patients with AIDS are particularly likely to be carnitine deficient.

Levocarnitine (L-carnitine) is a micronutrient found in meat and dairy products that plays a major role in energy metabolism. Preliminary research has shown that patients with end stage AIDS experienced decreased levels of fatigue after L-carnitine supplementation. This study will evaluate the effectiveness of L-carnitine to treat patients with carnitine deficiency, fatigue, and AIDS.

Participants in this study will be randomly assigned to receive either L-carnitine or placebo for 2 weeks. To reduce the possibility of side effects, the doses of L-carnitine and placebo will be titrated over 6 days to the desired study dose. After 2 weeks, participants receiving placebo will be switched over to receive L-carnitine. All participants will continue on L-carnitine for an additional 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* AIDS at Stage IV-C and estimated life expectancy < 6 months
* Karnofsky Performance Score > 50
* Clinically significant, persistent fatigue
* If undergoing pre-existing treatment for fatigue, must have been on a stable regimen for at least 4 weeks prior to study entry
* Concurrent use of epoetin alfa (PROCRIT®) will be allowed if the patient has been on a stable dose of epoetin alfa for at least 60 days prior to study entry

Exclusion Criteria:

* Severe cardiovascular, pulmonary, or renal function
* Hemodialysis
* Treatment or replacement therapy with any form of carnitine within 12 months prior to study entry
* Known sensitivity to carnitine
* Acute illness within 30 days of study entry that in the opinion of the study investigator would interfere with participation
* Active drug or alcohol use or dependence
* History of any central nervous system disease involving the brain that may put the patient at risk for seizure (e.g., primary or metastatic brain tumor, stroke) or history of seizure
* History of dementia, aphasia, or other deficits of cognition or speech/language function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2002-11; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Level of fatigue, measured by the fatigue sub-scale of the FAHI | Baseline; 2 weeks since starting L-carnitine or Placebo supplementation; 4 weeks (study termination)

SECONDARY OUTCOMES:
Changes in fatigue in the treatment and control groups | Baseline; 2 weeks since starting L-carnitine or Placebo supplementation; 4 weeks (study termination)
Changes in cognative status, mood, activity, and HGB levels mesured by BFI, LASA, KPS, and MSAS-SF | Baseline; 2 weeks since starting L-carnitine or Placebo supplementation; 4 weeks (study termination)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Cruciani, MD, PhD, Principal Investigator — Beth Israel Medical Center
Locations (1):
- Department of Pain Medicine and Palliative Care; Beth Israel Medical Center; First Avenue at 16th Street, New York, New York, United States